CLINICAL TRIAL: NCT00808496
Title: A Double Blind Randomized Controlled Trial to Compare Biannual Peripheral Magnetic Resonance Imaging, Radiography, and Standard of Care on Pharmacotherapeutic Escalation in Inflammatory Arthritis
Brief Title: The Effect of Biannual Monitoring With Magnetic Resonance Imaging (MRI), X-ray, or Usual Care on Treatment for Inflammatory Arthritis
Acronym: MRx
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ruben Tavares, PhD Candidate, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 200901
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Inflammatory Arthritis
Keywords: Magnetic resonance imaging; Radiography; Randomized controlled trial; Antirheumatic agents
MeSH Terms: conditions — Arthritis | interventions — X-Rays; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MRI (Experimental): Biannual disease progression monitoring with peripheral magnetic resonance imaging of the 2nd to 5th metacarpophalangeal joints of the worst-effected or dominant hand at baseline.
  Interventions: Other: MRI
- Radiography (Active Comparator): Biannual disease progression monitoring with radiography of both hands and wrists.
  Interventions: Other: Radiography
- Standard of Care (Placebo Comparator): Diagnostic imaging results (MRI or radiography) reported to upon requisition.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: MRI — Biannual disease progression monitoring with peripheral magnetic resonance imaging of the 2nd to 5th metacarpophalangeal joints of the worst-effected or dominant hand at baseline. Scored using the Xie-modified rheumatoid arthritis magnetic resonance imaging score (RAMRIS).
  MRI intervention group also undergoes radiography imaging. Only protocol determined smallest detectable changes on MRI reported.
  Other Names: Diagnostic imaging: 1T pMRI (OrthOne, ONI Medical Systems)
  Arms: MRI
Other: Radiography — Biannual disease progression monitoring with radiography of both hands and wrists. Scored using the van der Heijde-modified Sharp score.
  Radiography intervention group also undergoes MRI imaging. Only protocol determined smallest detectable changes on radiography reported.
  Other Names: Diagnostic Imaging: Conventional radiography.
  Arms: Radiography
Other: Standard of Care — Diagnostic imaging results (MRI or radiography) reported upon requisition. Standard of Care intervention group undergoes both MRI and radiography imaging. Upon requisition of either MRI or radiography, radiology reports are delivered as per institutional standard of care
  Other Names: Placebo control: see MRI and radiography interventions.
  Arms: Standard of Care

SUMMARY:
Inflammatory arthritis is a major cause of permanent joint damage. Joint damage causes functional disability and physical deformity. Many inflammatory arthritis patients develop permanent joint damage within the first two years of disease. Early, aggressive treatment with drugs called disease-modifying antirheumatic drugs (DMARDs) is known to reduce how quickly this damage occurs. Sometimes, however, even when patients' symptoms are under control, the disease continues to cause joint damage.

This study will determine if magnetic resonance imaging (also known as 'MRI') conducted every six months provides arthritis specialists with information to help them better treat peripheral inflammatory arthritis patients over the first two years of care. The effect of MRI will be compared to 1) the use of x-ray every six months; and, 2) the frequency at which these tests are usually used. The study will also determine if differences in treatment between the three groups result in differences in the well-being of patients.

A total of 186 patients with early signs of inflammatory arthritis will be studied. All participants will have an MRI and x-ray conducted every six months. One-third of participants (62 in total) will only have MRI information sent to their arthritis specialist (MRI group); 62 will have x-ray information sent (X-ray group); and, the remaining 62 will have x-ray information sent only when ordered by the arthritis specialist (Usual Care group). Negative disease progression reports will be sent to the arthritis specialist unless intervention allocation-specific disease progression is detected. In which case, a report blinded to imaging modality will be sent indicating the detection of disease progression relative to the last timepoint of progression, or baseline, as applicable. At any point in the study, the arthritis specialist can request a clinical MRI or x-ray for any participant.

Neither the participants nor their doctors will know to which group they are assigned. A computer program will randomly assign participants to one of the three groups using a technique called minimization. This technique accounts for differences between participants that are known to effect disease progression and treatment decisions. Using this technique, participants with similar disease will be evenly distributed between the three groups.

The results of this study will have a direct impact on care for new inflammatory arthritis patients. It will determine the benefits, if any, of regular monitoring of disease progression with MRI or x-ray. Using tests proven to help treatment decision-making, arthritis specialists will improve the care provided to new inflammatory arthritis patients.

DETAILED DESCRIPTION:
The proposed project is a double-blinded randomized-controlled trial to determine if biannual monitoring of inflammatory arthritis disease progression with 1.0T peripheral magnetic resonance imaging (pMRI) of the 2nd to 5th metacarpophalangeal joints of the worst-effected or dominant hand at baseline compared to conventional radiography of both hands and wrists, or standard of care, alters the frequency of pharmacological treatment escalation at two years. A sample size of 186 (62 per group) is required to determine mean differences in the rate of pharmacological treatment escalation between the three groups with 90% power at a 5% level of significance, assuming a 5% spontaneous remission rate, 15% missing data, and 5% annual attrition.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at study enrollment.
* At least three swollen joints; OR,
* Metacarpophalangeal joint(s) positive squeeze test; OR,
* Metatarsophalangeal joint(s) positive squeeze test; OR,
* At least 30 minutes of self-reported morning stiffness.
* At least six weeks of self-reported symptom duration.

Exclusion Criteria:

* Self-reported symptom onset prior to 17 years of age.
* Medical history of juvenile arthritis
* Evidence of viral arthritis
* A concomitant condition with medical priority over inflammatory arthritis, or that contraindicates treatment with DMARDs excluding sulfa allergy or medically controlled, non-terminal liver disease.
* Refusal to receive DMARD treatment
* Patients with a psychological deficit, or diminished capacity to provide independent, informed consent
* Any contraindication to MRI or x-ray
* Current or planned pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The frequency of antirheumatic treatment escalations. | Two years

SECONDARY OUTCOMES:
Change in van der Heijde-modified Sharp score of the hands and feet. | Two years
Change in 28-joint disease activity score (DAS28) | Two years
Change in health assessment questionnaire (HAQ) score | Two years
Change in Xie-modified rheumatoid arthritis magnetic resonance imaging score (RAMRIS) | Two years
Change in health utility index - mark 3 (HUI-III) | Two years
Change in EQ-5D | Two years
Number of smallest detectable changes | Two years
Change in the proportion of participants with radiography-determined erosions of the hands, wrists, or feet | Two years
Change in the number of radiography-determined erosions of the hands, wrists or feet | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Tavares, MBt MSc CCRA, Principal Investigator — McMaster University; Jonathan D Adachi, MD FRCPC, Study Chair — McMaster University; Maggie J Larche, MD PhD, Study Director — McMaster University; Colin E Webber, PhD CCPM, Study Director — McMaster University; Naveen Parasu, MD FRCPC, Study Director — McMaster University; Karen A Beattie, PhD, Study Director — McMaster University
Locations (1):
- McMaster University, Division of Rheumatology, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Brown AK, Conaghan PG, Karim Z, Quinn MA, Ikeda K, Peterfy CG, Hensor E, Wakefield RJ, O'Connor PJ, Emery P. An explanation for the apparent dissociation between clinical remission and continued structural deterioration in rheumatoid arthritis. Arthritis Rheum. 2008 Oct;58(10):2958-67. doi: 10.1002/art.23945. PMID 18821687
- [Background] Schiff MH, Hobbs KF, Gensler T, Keenan GF. A retrospective analysis of low-field strength magnetic resonance imaging and the management of patients with rheumatoid arthritis. Curr Med Res Opin. 2007 May;23(5):961-8. doi: 10.1185/030079907x178892. PMID 17519063
- [Background] McQueen FM, Stewart N, Crabbe J, Robinson E, Yeoman S, Tan PL, McLean L. Magnetic resonance imaging of the wrist in early rheumatoid arthritis reveals progression of erosions despite clinical improvement. Ann Rheum Dis. 1999 Mar;58(3):156-63. doi: 10.1136/ard.58.3.156. PMID 10364913
- [Background] Olech E, Freeston JE, Conaghan PG, Hensor EM, Emery P, Yocum D. Using extremity magnetic resonance imaging to assess and monitor early rheumatoid arthritis: the optimal joint combination to be scanned in clinical practice. J Rheumatol. 2008 Apr;35(4):580-3. Epub 2008 Mar 1. PMID 18322995
- [Background] Xie X, Webber CE, Adachi JD, O'Neill J, Inglis D, Bobba RS, Wu H. Quantitative, small bore, 1 Tesla, magnetic resonance imaging of the hands of patients with rheumatoid arthritis. Clin Exp Rheumatol. 2008 Sep-Oct;26(5):860-5. PMID 19032820
- [Background] van der Heijde DM, van Riel PL, Nuver-Zwart IH, Gribnau FW, vad de Putte LB. Effects of hydroxychloroquine and sulphasalazine on progression of joint damage in rheumatoid arthritis. Lancet. 1989 May 13;1(8646):1036-8. doi: 10.1016/s0140-6736(89)92442-2. PMID 2565997
- [Background] Taves DR. Minimization: a new method of assigning patients to treatment and control groups. Clin Pharmacol Ther. 1974 May;15(5):443-53. doi: 10.1002/cpt1974155443. No abstract available. PMID 4597226
- [Background] Saag KG, Teng GG, Patkar NM, Anuntiyo J, Finney C, Curtis JR, Paulus HE, Mudano A, Pisu M, Elkins-Melton M, Outman R, Allison JJ, Suarez Almazor M, Bridges SL Jr, Chatham WW, Hochberg M, MacLean C, Mikuls T, Moreland LW, O'Dell J, Turkiewicz AM, Furst DE; American College of Rheumatology. American College of Rheumatology 2008 recommendations for the use of nonbiologic and biologic disease-modifying antirheumatic drugs in rheumatoid arthritis. Arthritis Rheum. 2008 Jun 15;59(6):762-84. doi: 10.1002/art.23721. No abstract available. PMID 18512708
- [Background] Emery P, Breedveld FC, Dougados M, Kalden JR, Schiff MH, Smolen JS. Early referral recommendation for newly diagnosed rheumatoid arthritis: evidence based development of a clinical guide. Ann Rheum Dis. 2002 Apr;61(4):290-7. doi: 10.1136/ard.61.4.290. PMID 11874828
- [Derived] Tavares R, Beattie KA, Bensen WG, Bobba RS, Cividino AA, Finlay K, Goeree R, Hart LE, Jurriaans E, Larche MJ, Parasu N, Tarride JE, Webber CE, Adachi JD. A double-blind, randomized controlled trial to compare the effect of biannual peripheral magnetic resonance imaging, radiography and standard of care disease progression monitoring on pharmacotherapeutic escalation in rheumatoid and undifferentiated inflammatory arthritis: study protocol for a randomized controlled trial. Trials. 2014 Jul 5;15:268. doi: 10.1186/1745-6215-15-268. PMID 24997587